CLINICAL TRIAL: NCT05347732
Title: Predictors of Failed Thrombolysis in Acute ST-segment Elevation Myocardial Infarction
Brief Title: Predictors of Failed Thrombolysis in Acute Myocardial Infarction
Acronym: TROFAMI
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ragnhild Helseth, Cardiologist, PhD, Oslo University Hospital
Other Study IDs: 341357
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Successfull thrombolysis — Biomarker levels will be compared between patients with successful and failed thrombolysis.

SUMMARY:
The purpose of this observational study is to assess why thrombolytic treatment with tissue-plasminogen activator (t-PA) fails in patients with acute ST-segment elevation myocardial infarction (STEMI). The study will include 200 STEMI patients at the time of arrival at Oslo University Hospital Ullevål after receiving prehospital thrombolysis. A blood sample will be taken immediately for the study of factors related to coagulation, fibrinolysis and inflammation. Levels of the biomarkers will be compared between patients with successful and failed thrombolysis.

DETAILED DESCRIPTION:
This study aims to explore why thrombolytic treatment with tissue-plasminogen activator (t-PA) fails in up to 50 % of pasients with acute ST-segment elevation myocardial infarction (STEMI). This is important in Norway due to the long geographic distances and the fact that up to 70 % of STEMI patients in some Norwegian areas receive thrombolysis in stead of primary, invasive revascularization with percutaneous coronary intervention (PCI). Today, no well-defined biomarker or score can predict the successfulness of thrombolytic therapy during STEMI. As failed thrombolysis leads to larger myocardial infarctions and poorer outcome, defining factors for improved risk stratification is important.

The TROFAMI study is a prospective study which will include 200 STEMI patients given prehospital thrombolysis. A blood sample will be taken immediately after hospital admission for the analysis of potential relevant biomarkers related to coagulation, fibrinolysis and inflammation. The biomarkers will be evaluated against the successfullness or not of thrombolysis.

Oslo University Hospital is the largest STEMI center in Norway. Each year, approximately 100 STEMI patients given prehospital thrombolysis are hospitalized at Ullevål. The inclusion is anticipated to take place during the time period 2022-2024.

ELIGIBILITY:
Inclusion Criteria:

STEMI patients > 18 years given prehospital thrombolysis.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all STEM patients who have received prehospital thrombolysis before hospital admission.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2035-01-03 (Estimated)

PRIMARY OUTCOMES:
Failed thrombolysis | Decided immediately after hospital admission.
  Persistent chest pain and/or < 50 % ST segment resolution

CONTACTS AND LOCATIONS:
Overall Officials: Ragnhild Helseth, MD PhD, Study Director — Department of Cardiology, Oslo University Hospital Ullevål
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No